CLINICAL TRIAL: NCT06215170
Title: SafeMedWaste At-Home, Environmentally-Friendly Opioid Disposal Kit for Orthopedic Post-Operative Surgical Patients to Reduce Opioids Available for Diversion
Acronym: Drug Disposal
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SafeMedWaste, Inc. (Industry)
Collaborators: Prisma Health-Midlands (Other); University of South Carolina (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SafeMedWasteCT2023; 1R43DA057750-01A1 (NIH)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; Drug Disposal; at-home drug disposal; Drug Diversion; Opioid Disposal
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): General Instructions on Opioid Disposal
- Treatment (Active Comparator): General Instructions on opioid disposal Device: SafeMedWaste Opioid Disposal Kit
  Interventions: Device: SafeMedWaste

INTERVENTIONS:
Device: SafeMedWaste — SafeMedWaste opioid disposal kit
  Arms: Treatment

SUMMARY:
There is an urgent unmet medical need for a cost-effective, environmentally friendly, in-home opioid disposal solution for surgical patients that is clinically proven to reduce opioid use disorder that is substantiated with economic data. SafeMedWaste, Inc. (SMW) has developed the patented SafeMedWaste in-home drug disposal container, that completely destroys opioids within minutes and can be placed in the regular trash, without risk of ground or municipal water contamination.

A pilot randomized clinical trial will evaluate the use of SafeMedWaste in 300 adult patients in outpatient surgery clinics undergoing shoulder and knee surgery.

DETAILED DESCRIPTION:
The trial will evaluate opioid disposal rates and events related to opioid diversion and use disorder in 300 adult patients 18 years of age and older undergoing outpatient knee and shoulder surgery who are prescribed opioids to manage their acute post-surgical pain.

Patients will be randomized into two arms. During the standard of care post op visits (2-, 6- and 10- weeks), when the treating physician has determined that the patient will no longer need opioids to manage their post-surgical pain, all patients will receive general instructions by video on opioid disposal recorded by one of the orthopedic surgeons. Patients in the treatment arm will also be given the SafeMedWaste opioid disposal system and watch an instructional video on how to use the product.

All patients will complete a pre-surgery survey and a post-surgery survey 90 days after surgery. Patients will self-report their disposal or non-disposal of the drugs, documented with pictures uploaded to the patient's MyChart account. Data from the surveys will be statistically analyzed to identify significant factors that influenced patients' behavior vis-à-vis opioid disposal.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Subject is 18 + years of age
  * Subject is opioid naive (within the last 3 months), as evidenced by MyChart patient record or response to medical history questions
  * Subject is scheduled to undergo shoulder and/or knee surgery

Exclusion Criteria:

* Subject has a history of opioid addiction, as evidenced by MyChart patient record or response to medical history questions
* Subject is currently utilizing prescription narcotics for any reason, as evidenced by MyChart patient record or response to medical history questions
* Subject does not have the mental capacity to make their own healthcare decisions
* Subject is unable to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Opioid disposal compliance | Within 3 months following surgery
  Opioid disposal compliance will be tracked up to 3 months post-surgery, as reported by patients in post-surgery survey and/or documented with pictures uploaded by patient to MyChart.

OTHER OUTCOMES:
Reasons for disposal/non- disposal | Within 3 months following surgery
  Reasons why the patient chose to dispose of opioids or chose not to, as reported in the post- surgery survey, will be statistically analyzed and correlated as appropriate to other data.
Time of disposal | Within 3 months following surgery
  When the patients dispose of opioids, as reported by patients in post-surgery survey and/or documented with pictures in MyChart, will be tracked up to 3 months post-surgery.
Amount of opioids used | Within 3 months following surgery
  The amount of opioids used will be tracked at visit weeks 2, 6 and 10, post surgery, through clinic pill counts, or as self-reported by patients up to 3 months.
Opioid Use Disorder (OUD) | Within 3 months following surgery
  Any OUD reported in the patient medical record will be tracked up to 3 months following surgery.
Diversion event | Within 3 months following surgery
  Any diversion event as described by patient at clinical visit or in post-surgery survey will be recorded.
Pre-Surgery Survey | At enrollment
  Pre-Surgery Survey, see Ex. 1, Protection of Human Subjects, will be completed by patients at enrollment. Questions include patient past surgical experience and attitudes toward pain. Data will be recorded in REDCap and statistically analyzed.
Post-Surgery Survey | 3 months following surgery
  Patients will answer post-surgery survey, see Ex. 2, Protection of Human Subjects, within 3 months following surgery. Questions include pain experiences from their surgery and disposal compliance. Data will be recorded in REDCAP and statistically analyzed for correlations of patient attitudes toward and experience with pain and other factors to disposal compliance to create clinician/patient education protocols to be studied in future trial.
Provider Satisfaction Survey | Upon study completion
  Provider participants will answer Provider Satisfaction survey, see Ex. 4, Protection of Human Subjects, upon study completion. Data will be recorded in REDCap and statistically analyzed.

IPD SHARING:
Plan to Share IPD: Undecided